CLINICAL TRIAL: NCT06699069
Title: The Effect of Exercise on Serum Irisin Levels in Hypothyroid Sprague Dawley Rats
Brief Title: Effect of Exercise on Irisin Levels of Hypothyroid Rats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRC/20/232 Fatima Iqbal
Record Dates: First submitted 2021-02-02; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Hypothyroidism
Keywords: Exercise; Irisin; Hypothyroidism
MeSH Terms: conditions — Hypothyroidism; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Control or Euthyroid) total number of rats=20 (Experimental): Fed on normal standard diet
  Interventions: Other: Control or Euthyroid group
- Group II (Hypothyroid) total number of rats=20 (Experimental): Experimental hypothyroidism will be induced by administration of propylthiouracil for three weeks in the form of tablets diluted in water
  Interventions: Other: Hypothyroid group
- Group III (Hypothyroid received exercise) total number of rats=20 (Experimental): Rats will be subjected to chronic swimming. The swimming protocol will consist of 8 weeks of low-intensity swimming exercise.
  Interventions: Other: Hypothyroid group received exercise

INTERVENTIONS:
Other: Control or Euthyroid group — Fed on normal standard diet
  Arms: Group I (Control or Euthyroid) total number of rats=20
Other: Hypothyroid group — Experimental hypothyroidism will be induced by administration of propylthiouracil for three weeks in the form of tablets diluted in water
  Arms: Group II (Hypothyroid) total number of rats=20
Other: Hypothyroid group received exercise — Rats will be subjected to chronic swimming. The swimming protocol will consist of 8 weeks of low-intensity swimming exercise. The exercise groups will be adapted to a round water tank (70 cm × 70 cm) containing water at 28 ± 2°C for 3 days (10-45 min/day). The rats will then begin swimming, 45 min/day for the first two weeks at 10am and 60 min/day for the last six weeks at 10am
  Arms: Group III (Hypothyroid received exercise) total number of rats=20

SUMMARY:
The aim of study was to evaluate the role of exercise on serum irisin levels in hypothyroid rats.

DETAILED DESCRIPTION:
Contracting skeletal muscle acts as an endocrine organ, capable of secreting hormones called myokines, such as interleukin 1, Interleukin 15 and Irisin. Myokines are important for regulation of glucose and lipid metabolism. Among these, irisin, is an exercise induced polypeptide, secreted mainly by skeletal muscles and adipose tissue. Irisin is also secreted in small amounts from cardiac muscle, pancreas and sebaceous glands. It is cleaved and secreted from fibronectin type III domain-containing protein 5 (FNDC5 gene) and is regulated by the peroxisome proliferator-activated receptor-γ co activator 1-α (PGC1-α) .

The most important function of Irisin is thermogenesis, by inducing the browning of white adipose tissue, thereby increasing energy consumption, encouraging weight loss and decreasing dietary insulin resistance. Linking Irisin levels with obesity, its mechanism shows that after exercise there is up regulation of a thermogenin ,an Uncoupling Protein-1 (UCP-1) Thyroid hormone also plays an important role in glucose-lipid metabolism and energy homeostasis. Hypothyroidism, a decrease in thyroid hormone levels, can lead to obesity and metabolic syndrome. It has been found that thyroid hormone is also involved in thermogenesis by inducing browning of white adipose tissue, through thyroid hormone receptors. In hypothyroidism, many metabolic processes in the body are affected such as differentiation in the adipose tissue. Increased thyroid stimulating hormone (TSH) causes adipogenesis by stimulating pre-adipocyte differentiation directly through the receptors in the adipose tissue . Fatty tissue is increased by adipocyte hypertrophy as a consequence of previous adipogenesis, and newly formed adipocyte-8, resulting in clinical obesity.

FNDC5 (Fibronectin type III domain-containing protein 5), which is the precursor of irisin, is a protein that is encoded by the FNDC5 gene, is present in many tissues, including the thyroid tissue and therefore effects thyroid hormone.

Dysregulation of both Thyroid and Irisin hormones result in metabolic syndrome. The metabolic syndrome is a common metabolic disorder that has been linked to the increasing prevalence of obesity. By regulating thyroid hormone levels, irisin has a powerful impact on metabolism and thermogenesis. The association of irisin with the thyroid hormone in hypothyroidism still remains unknown and is controversial, and requires further confirmatory studies on experimental models.

Regular exercise is known to have significant beneficial effects on the metabolic health and this is mediated by skeletal muscle. Contracting skeletal muscle is the source of Irisin. Studies have shown an increase in post exercise Irisin levels

ELIGIBILITY:
Inclusion Criteria:

* Male adult rats weighing approx. 200-250gms
* 6 to 8 week old rats

Exclusion Criteria:

* Female rats will be excluded.
* Rats with any obvious pathology
* The rats weighing >200gm

Ages: 6 Weeks to 8 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male Sprague Dawley Rats
Enrollment: 30 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Serum Triiodothyronine T3 | 11th week
  Estimation of serum free triiodothyronine (FT3) levels (ng/ml) by radioimmunoassay
Serum Thyroxine | 11th week
  Estimation of serum free thyroxin (FT4) levels (μg/dl) by radioimmunoassay
Serum Irisin | 11th week
  Estimation of serum irisin levels (μg/ml) by using enzyme - linked immunosorbent assay (ELISA) using irisin competitive ELISA Kit
Serum Thyroid Stimulating Hormone | 11th week
  By radioimmunoassay
Serum Triglycerides (TG) | 11th week
  By enzymatic method using micro lab analyzer
Serum High Density Lipoproteins (HDL) | 11th week
  Determined by precipitating method using micro lab analyzer
Serum Low Density Lipoproteins (LDL) | 11th week
  LDL= Total cholesterol-HDL-TG/5

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Ali, PhD, Principal Investigator — Riphah International University
Locations (1):
- National Institute of Health, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez Munoz IY, Camarillo Romero EDS, Garduno Garcia JJ. Irisin a Novel Metabolic Biomarker: Present Knowledge and Future Directions. Int J Endocrinol. 2018 Oct 9;2018:7816806. doi: 10.1155/2018/7816806. eCollection 2018. PMID 30402097
- [Background] Korta P, Pochec E, Mazur-Bialy A. Irisin as a Multifunctional Protein: Implications for Health and Certain Diseases. Medicina (Kaunas). 2019 Aug 15;55(8):485. doi: 10.3390/medicina55080485. PMID 31443222
- [Background] Gizaw M, Anandakumar P, Debela T. A Review on the Role of Irisin in Insulin Resistance and Type 2 Diabetes Mellitus. J Pharmacopuncture. 2017 Dec;20(4):235-242. doi: 10.3831/KPI.2017.20.029. Epub 2017 Oct 10. PMID 30151293 (Retraction: PMID 32322435 J Pharmacopuncture. 2020 Mar 31;23(1):42-43)
- [Background] Uc ZA, Gorar S, Mizrak S, Gullu S. Irisin levels increase after treatment in patients with newly diagnosed Hashimoto thyroiditis. J Endocrinol Invest. 2019 Feb;42(2):175-181. doi: 10.1007/s40618-018-0899-8. Epub 2018 May 18. PMID 29777516
- [Background] Maalouf GE, El Khoury D. Exercise-Induced Irisin, the Fat Browning Myokine, as a Potential Anticancer Agent. J Obes. 2019 Apr 1;2019:6561726. doi: 10.1155/2019/6561726. eCollection 2019. PMID 31065382
- [Background] Deshmukh V, Farishta F, Bhole M. Thyroid Dysfunction in Patients with Metabolic Syndrome: A Cross-Sectional, Epidemiological, Pan-India Study. Int J Endocrinol. 2018 Dec 25;2018:2930251. doi: 10.1155/2018/2930251. eCollection 2018. PMID 30675157
- [Background] Abdel Moety DA. Evaluation of Serum Irisin and Creatine Kinase Levels in Hypo- and Hyperthyroid Rats. Al-Azhar Med J. 2017;46(1):163-74.
- [Background] Ates I, Altay M, Topcuoglu C, Yilmaz FM. Circulating levels of irisin is elevated in hypothyroidism, a case-control study. Arch Endocrinol Metab. 2016 Apr;60(2):95-100. doi: 10.1590/2359-3997000000077. Epub 2015 Jul 21. PMID 26201007
- [Background] Yang N, Zhang H, Gao X, Miao L, Yao Z, Xu Y, Wang G. Role of irisin in Chinese patients with hypothyroidism: an interventional study. J Int Med Res. 2019 Apr;47(4):1592-1601. doi: 10.1177/0300060518824445. Epub 2019 Feb 6. PMID 30722716
- [Background] Rochlani Y, Pothineni NV, Kovelamudi S, Mehta JL. Metabolic syndrome: pathophysiology, management, and modulation by natural compounds. Ther Adv Cardiovasc Dis. 2017 Aug;11(8):215-225. doi: 10.1177/1753944717711379. Epub 2017 Jun 22. PMID 28639538
- [Background] Teixeira PFDS, Dos Santos PB, Pazos-Moura CC. The role of thyroid hormone in metabolism and metabolic syndrome. Ther Adv Endocrinol Metab. 2020 May 13;11:2042018820917869. doi: 10.1177/2042018820917869. eCollection 2020. PMID 32489580
- [Background] Kurdiova T, Balaz M, Vician M, Maderova D, Vlcek M, Valkovic L, Srbecky M, Imrich R, Kyselovicova O, Belan V, Jelok I, Wolfrum C, Klimes I, Krssak M, Zemkova E, Gasperikova D, Ukropec J, Ukropcova B. Effects of obesity, diabetes and exercise on Fndc5 gene expression and irisin release in human skeletal muscle and adipose tissue: in vivo and in vitro studies. J Physiol. 2014 Mar 1;592(5):1091-107. doi: 10.1113/jphysiol.2013.264655. Epub 2013 Dec 2. PMID 24297848